CLINICAL TRIAL: NCT04696614
Title: Developing and Testing the Effect of Exercise Intervention Using a SMART Design on Reducing Visceral Adipose Tissue in Community Residents: A Mixed-Method, Longitudinal Study.
Brief Title: Testing the Effect of Exercise Intervention Using a SMART Design.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Chang, Principal Investigator, National Taiwan University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 108466
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Fat Burn
Keywords: sequential multiple assignment randomized trial; exercise; visceral adipose tissue
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with 1:1 equal allocation at baseline to one of two first-stage interventions (8 weeks aerobic exercise (AE) or interval training). Those who exhibit early signs of nonresponse determined by a tailoring variable (reduced (visceral adipose tissue (VAT) < 3%) will then be rerandomized to one of two second-stage interventions (AE + RE (resistance exercise) vs interval training or AE), also with 1:1 equal allocation, whereas those who have a significant response to the first-stage intervention will continue to receive the same exercise treatment until 16 weeks.
Who Masked: Outcomes Assessor
Masking Description: singal blinding for the assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- aerobic exercise to aerobic exercise (Experimental): first 8-week: aerobic exercise second 8-week: aerobic exercise
  Interventions: Behavioral: exercise
- aerobic exercise to interval training (Experimental): first 8-week: aerobic exercise second 8-week: interval training
  Interventions: Behavioral: exercise
- aerobic exercise to aerobic exercise +resistance exercise (Experimental): first 8-week: aerobic exercise second 8-week: aerobic exercise +resistance exercise
  Interventions: Behavioral: exercise
- interval training to interval training (Experimental): first 8-week: interval training second 8-week: interval training
  Interventions: Behavioral: exercise
- interval training to aerobic exercise (Experimental): first 8-week: interval training second 8-week: aerobic exercise
  Interventions: Behavioral: exercise
- interval training to aerobic exercise+resistance exercise (Experimental): first 8-week: interval training second 8-week: aerobic exercise +resistance exercise
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — intervention groups provided different sequential modality of exercise

SUMMARY:
Exercise is the most effective way on reducing visceral adipose tissue (VAT), which is strongly linked with obesity to hypertension, cardiovascular disease, and insulin resistance. However, the current exercise dosage for reducing VAT cannot be accurately quantified. The aims of this study are to develop and test the optimal exercise dosage and sequence for reducing VAT in overweight and obese community residents. Purposive sampling will be used to enroll at least 206 participants aged 40-65 years and body fat more than 30% without diet control from 2 community centers in southern Taiwan. The project will use the sequential multiple assignment randomized trial (SMART) design to conduct a 16-week 2-stage (each for 8-weeks) adaptive exercise intervention for community residents. In the first stage, participants will be randomized into groups performing 8 weeks either moderate intensity of aerobic exercise or interval training 3 times per week. Participants whose VAT does not decrease by over 3%, measured using a body composition analyzer, compared with the baseline will be 1:1 rerandomized into groups with aerobic exercise combined with resistance exercise or received the exchange of first stage treatment (interval training or aerobic exercise) in the second stage. Those with substantial response to the first-stage intervention (VAT reduction of more than 3%) will continue to receive the same exercise treatment until 16 weeks. Linear mixed model, weighted and replicated regression will be used to identify the optimal sequence of exercises for the greatest reduction in VAT. The findings can assist clinical health workers to develop exercise prescriptions for effectively reducing VAT, and help community residents reduce VAT through exercise to achieve the health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Community residents (a) who are 40-65 years old without diet control, (b) body fat ≧ 30% measured by body composition analyzer, and (c) can communicate in Mandarin or Taiwanese will be included.

Exclusion Criteria:

* This study will exclude residents with (a) recent unstable condition involving stroke or those with heart disease, handicap, pregnancy, mental disorders, systolic BP > 200 mmHg, or diastolic BP >110 mmHg; and (b) those with contraindications in body composition analyzer measurement including people with pacemakers, artificial metal joints, amputated hands or feet, and those who cannot be cooperated with standing during testing.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
visceral adipose tissue | three times (baseline, change visceral adipose tissue from Baseline to 8 week, change visceral adipose tissue from Baseline to 16 week)
  measured using body composition analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Community Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang YH, Lee YH, Wu KL, Hsu WL, Hung H, Shun SC. Exercise Strategy for Reducing Visceral Adipose Tissue in Community Residents With Obesity: A Sequential Multiple Assignment Randomized Trial. J Nurs Res. 2025 Apr 1;33(2):e385. doi: 10.1097/jnr.0000000000000662. PMID 40019278